CLINICAL TRIAL: NCT02556684
Title: A Prospective Study to Evaluate Dynamic Breast-Specific Gamma Imaging in Monitoring Tumor Responses in Patients With Locally Advanced Breast Cancer Undergoing Neoadjuvant Chemotherapy
Brief Title: Breast-Specific Gamma Imaging and Locally Advanced Breast Cancer Undergoing Neoadjuvant Chemotherapy
Acronym: BSGILAB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Zhejiang University (Other)
Responsible Party: Principal Investigator, Zhigang Zhang, Dr, Zhejiang University
Other Study IDs: BSGILAB001
Record Dates: First submitted 2015-09-11; First posted 2015-09-22 (Estimated); Last update posted 2019-04-11 (Actual); Status verified 2019-04

CONDITIONS: Breast Cancer
Keywords: Breast-Specific Gamma Imaging; Locally Advanced Breast Cancer; Neoadjuvant Chemotherapy; BSGI
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

SUMMARY:
A prospective cohort study design will be conducted. Patients with LABC who receive chemotherapy will undergo physical examination, ultrasound, MRI, and BSGI at baseline, midway, and at the completion of chemotherapy. Approximately 100 patients will be recruited over a 2-year period. This study will give clinicians further insight into the usefulness of ultrasound, MRI, and BSGI in monitoring treatment responses in patients with LABC. This could potentially lead to changes in clinical management of these patients.

DETAILED DESCRIPTION:
Locally advanced breast cancer (LABC) is usually treated with neoadjuvant chemotherapy followed by surgery. At present, monitoring of tumor responses to chemotherapy is primarily carried out using physical examination at the beginning of each chemotherapy cycle. Differentiating viable tumor tissue from inflammation or fibrotic scar tissue can be difficult. There is a growing body of evidence that newer imaging techniques such as positron emission tomography (PET) and magnetic resonance imaging (MRI) may be better at determining whether or not the tumor is actually shrinking, but their sensitivity and specificity were not ideal. Breast-specific gamma imaging (BSGI) using 99mTcsestamibi is a relatively new nuclear medicine imaging technique for breast tumor detection. BSGI shows higher sensitivity than conventional scintimammography in the detection of small breast cancer lesions owing to its high resolution. BSGI is a useful complementary tool to ultrasound, mammography and MRI in breast cancer diagnosis, especially in dense breasts and multifocal or multicentric disease; however, little is known about the ability of BSGI to predict of clinical and pathological response to neo-adjuvant chemotherapy in patients with locally advanced breast cancer. The purpose of this study is to determine the sensitivity and specificity of BSGI in evaluating tumor responses to chemotherapy in patients with LABC and compare this with physical examination, ultrasound, mammography and MRI, which is the current conventional standard of care. A prospective cohort study design will be conducted. Patients with LABC who receive chemotherapy will undergo physical examination, ultrasound, MRI, and BSGI at baseline, midway, and at the completion of chemotherapy. Approximately 100 patients will be recruited over a 2-year period. This study will give clinicians further insight into the usefulness of ultrasound, MRI, and BSGI in monitoring treatment responses in patients with LABC. This could potentially lead to changes in clinical management of these patients.

ELIGIBILITY:
Inclusion Criteria

* 18 Years and older, and histologic proof of breast cancer (invasive ductal or lobular carcinoma-not breast sarcoma or lymphoma)
* Patients having a clinical diagnosis of locally advanced breast cancer (T3 or T4, or N2 according to TNM classification) including inflammatory breast cancer.
* Patients must be able to undergo neoadjuvant chemotherapy.
* Eastern Cooperative Oncology Group (ECOG) performance status of 0, 1 or 2 sufficient to undergo chemotherapy

Exclusion Criteria

* Previously treated cancer other than non melanotic skin cancer or carcinoma in situ of the cervix, unless disease-free for 5 years or greater.
* Evidence of metastatic disease (found on chest X-ray, liver ultrasound or bone scan).
* Previous chemotherapy or hormonal therapy for breast cancer.
* Active infection or other significant illnesses which could hamper their ability to tolerate chemotherapy
* Significant concurrent medical problems (e.g. uncontrolled diabetes, active cardiac disease, severe chronic obstructive pulmonary disease) making the patient unfit for surgery.
* Any condition that could interfere with their ability to provide informed consent such as dementia or severe cognitive impairment.
* Pregnant or lactating females.
* Inadequate hematologic, renal and liver function as measured by CBC (WBC<4.0 x 109, Hb<100 g/L, plt count<100 x 109), and abnormal hepatic transaminases (AST, ALT, GGT, alkaline phosphatase>2x normal), elevated total bilirubin, and elevated serum creatinine (Cr>110 micromol/L).
* Any contraindication to undergoing MRI or BSGI.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Locally Advanced Breast Cancer Undergoing Neoadjuvant Chemotherapy
Sampling Method: Probability Sample
Enrollment: 200 (Estimated)
Dates: Start 2015-09 (Actual); Primary Completion 2020-10 (Estimated); Study Completion 2020-10 (Estimated)

PRIMARY OUTCOMES:
Sensitivity/Specificity | 2 YEARS
  BSGI have a high sensitivity/specificity t in predicting which LABC patients achieve a complete pathologic response (pCR) following neo-adjuvant chemotherapy

SECONDARY OUTCOMES:
pathologic complete response | 2 YEARS
  BSCGI might changes in clinical management by identifying non-responders earlier than with other examinations.
Overall Survival | 2 YEARS
  BSGI predict long-term survival

CONTACTS AND LOCATIONS:
Overall Officials: Jian Huang, Dr, Study Chair — Second Affiliated Hospital of Zhejiang University School of Medicine
Locations (1):
- Cancer institute, Hangzhou, Zhejiang, China

REFERENCES:
- [Background] Gong Z, Williams MB. Comparison of breast specific gamma imaging and molecular breast tomosynthesis in breast cancer detection: Evaluation in phantoms. Med Phys. 2015 Jul;42(7):4250-9. doi: 10.1118/1.4922398. PMID 26133623
- [Background] Kelley KA, Crawford JD, Thomas K, Gardiner SK, Johnson NG. A Comparison of Breast-Specific Gamma Imaging of Invasive Lobular Carcinomas and Ductal Carcinomas. JAMA Surg. 2015 Aug;150(8):816-8. doi: 10.1001/jamasurg.2015.0965. No abstract available. PMID 26107618
- [Background] Yoon HJ, Kim Y, Chang KT, Kim BS. Prognostic value of semi-quantitative tumor uptake on Tc-99m sestamibi breast-specific gamma imaging in invasive ductal breast cancer. Ann Nucl Med. 2015 Aug;29(7):553-60. doi: 10.1007/s12149-015-0977-3. Epub 2015 May 5. PMID 25939640
- [Background] Lee HS, Ko BS, Ahn SH, Son BH, Lee JW, Kim HJ, Yu JH, Kim SB, Jung KH, Ahn JH, Cha JH, Kim HH, Lee HJ, Song IH, Gong G, Park SH, Lee JJ, Moon DH. Diagnostic performance of breast-specific gamma imaging in the assessment of residual tumor after neoadjuvant chemotherapy in breast cancer patients. Breast Cancer Res Treat. 2014 May;145(1):91-100. doi: 10.1007/s10549-014-2920-z. Epub 2014 Mar 27. PMID 24671359
- [Background] Sun Y, Wei W, Yang HW, Liu JL. Clinical usefulness of breast-specific gamma imaging as an adjunct modality to mammography for diagnosis of breast cancer: a systemic review and meta-analysis. Eur J Nucl Med Mol Imaging. 2013 Feb;40(3):450-63. doi: 10.1007/s00259-012-2279-5. Epub 2012 Nov 14. PMID 23151912